CLINICAL TRIAL: NCT04793646
Title: Prospective Randomized, Double-blind Controlled Clinical Study of N-acetylcysteine for Treatment of Dryness Symptoms Due to Primary Sjogren's Syndrome
Brief Title: N-acetylcysteine for Primary Sjögren's Syndrome
Acronym: NACSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24088719.4.0000.0068
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Sjögren Syndrome; Sicca Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind controlled study of N-acetylcysteine for treatment of dryness symptoms due to primary Sjogren's syndrome
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding of identical bottles of N-acetylcysteine and placebo syrup
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcysteine syrup (Active Comparator): Thirty pSS patients
  Interventions: Drug: N-acetylcysteine syrup
- Placebo syrup (Placebo Comparator): Thirty pSS patients
  Interventions: Drug: Placebo syrup

INTERVENTIONS:
Drug: N-acetylcysteine syrup — N-acetylcysteine syrup 600 mg (15 mL) twice a day for 3 months
  Other Names: N-acetylcysteine
  Arms: N-acetylcysteine syrup
Drug: Placebo syrup — Placebo syrup 15 mL twice a day for 3 months
  Other Names: Placebo
  Arms: Placebo syrup

SUMMARY:
N-acetylcysteine (NAC) allows the elimination of reactive oxygen species (ROSs) and it has an anti-inflammatory effect. For this reason, NAC has been used and researched for treatment of several diseases, such as autoimmune diseases. In these diseases there are a process of oxidative stress due to chronic inflammation, which promotes an imbalance between ROSs levels and the cellular capacity to eliminate reactive intermediates and repair the resulting damage through antioxidants. The imbalance between the production of free radicals from oxygen and antioxidant species may also be involved in the pathogenesis of primary Sjögren's syndrome (pSS). In fact, increased levels of oxidative stress markers were detected in biopsy samples from minor salivary glands in these patients. Treatment of pSS is not well established and it is also not able to modify the evolution of the disease, being often only symptomatic. In addition, there is little data in the literature regarding the true efficacy of NAC in the treatment of pSS and the few existing studies have evaluated heterogeneous populations (including patients with other causes of sicca syndrome) and validated instruments to measure the symptom index and disease activity were not use in these previous studies. Thus, the present randomized double-blind clinical study aims to evaluate the efficacy of NAC in the control of sicca syndrome symptoms in a homogeneous population of patients with pSS (not only regarding the classification criteria, but also regarding the low rate of systemic disease activity at study inclusion) through tests widely accepted in the literature. Additionally, the investigators will study the possible role of NAC on oxidative stress in peripheral blood and saliva of these patients.

DETAILED DESCRIPTION:
Study design: This is a prospective, randomized, double-blind controlled study of N-acetylcysteine (600 mg orally every 12 hours in the form of syrup) lasting 12 weeks for the treatment of sicca syndrome symptoms due to pSS.

Patients: Sixty adult female patients (aged >=18 years), with a well-established diagnosis of pSS (2016 American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) and/or 2002 American-European Consensus classification criteria) and follow-up regularly at the Sjögren Syndrome Outpatient Clinic of the Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HCFMUSP).

Sample size: There is only a controlled study of NAC for treatment of SS, which included a heterogeneous population with a total of 26 patients and who observed superiority to placebo in the sicca symptoms control. Based on this study, the investigators will work with a convenience sample of 60 patients.

Clinical evaluation: It will be carried out at study inclusion, 4 weeks and 12 weeks through clinical instruments widely accepted in the literature.

Laboratorial evaluation: ROs will also be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the study according to signed informed consent.
* Filling the pSS classification criteria.
* Absence of other autoimmune associates systemic diseases.
* EULAR Sjögren Syndrome Disease Activity Index (ESSDAI) <= 5.
* Prednisone dose < 20 mg/day at study inclusion.
* Without pilocarpine or cevimeline use at study inclusion.
* No use of N-acetylcysteine for at least 1 month before study inclusion.

Exclusion Criteria:

* Diabetes, sarcoidosis, previous history of head and neck radiotherapy or iodine therapy, positive serologies for HIV, hepatitis B and C, graft versus host disease, IgG4 (immunoglobulin G4) related disease, and current use of antidepressants tricyclics.
* Current use of biological therapy.
* Current smoking.
* Alcoholism.
* Liver cirrhosis and chronic kidney disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) | 3 months
  Comparative analysis of ESSPRI values

SECONDARY OUTCOMES:
Xerostomia inventory | 3 months
  Comparative analysis of xerostomia inventory values

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Pasoto, MD, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (2):
- Brazil (2):
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vitali C, Bombardieri S, Jonsson R, Moutsopoulos HM, Alexander EL, Carsons SE, Daniels TE, Fox PC, Fox RI, Kassan SS, Pillemer SR, Talal N, Weisman MH; European Study Group on Classification Criteria for Sjogren's Syndrome. Classification criteria for Sjogren's syndrome: a revised version of the European criteria proposed by the American-European Consensus Group. Ann Rheum Dis. 2002 Jun;61(6):554-8. doi: 10.1136/ard.61.6.554. PMID 12006334
- [Background] Shiboski CH, Shiboski SC, Seror R, Criswell LA, Labetoulle M, Lietman TM, Rasmussen A, Scofield H, Vitali C, Bowman SJ, Mariette X; International Sjogren's Syndrome Criteria Working Group. 2016 American College of Rheumatology/European League Against Rheumatism classification criteria for primary Sjogren's syndrome: A consensus and data-driven methodology involving three international patient cohorts. Ann Rheum Dis. 2017 Jan;76(1):9-16. doi: 10.1136/annrheumdis-2016-210571. Epub 2016 Oct 26. PMID 27789466
- [Background] Seror R, Ravaud P, Mariette X, Bootsma H, Theander E, Hansen A, Ramos-Casals M, Dorner T, Bombardieri S, Hachulla E, Brun JG, Kruize AA, Praprotnik S, Tomsic M, Gottenberg JE, Devauchelle V, Devita S, Vollenweider C, Mandl T, Tzioufas A, Carsons S, Saraux A, Sutcliffe N, Vitali C, Bowman SJ; EULAR Sjogren's Task Force. EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI): development of a consensus patient index for primary Sjogren's syndrome. Ann Rheum Dis. 2011 Jun;70(6):968-72. doi: 10.1136/ard.2010.143743. Epub 2011 Feb 22. PMID 21345815
- [Background] Seror R, Ravaud P, Bowman SJ, Baron G, Tzioufas A, Theander E, Gottenberg JE, Bootsma H, Mariette X, Vitali C; EULAR Sjogren's Task Force. EULAR Sjogren's syndrome disease activity index: development of a consensus systemic disease activity index for primary Sjogren's syndrome. Ann Rheum Dis. 2010 Jun;69(6):1103-9. doi: 10.1136/ard.2009.110619. Epub 2009 Jun 28. PMID 19561361
- [Background] Walters MT, Rubin CE, Keightley SJ, Ward CD, Cawley MI. A double-blind, cross-over, study of oral N-acetylcysteine in Sjogren's syndrome. Scand J Rheumatol Suppl. 1986;61:253-8. PMID 3296153
- [Background] Ramos-Casals M, Brito-Zeron P, Siso-Almirall A, Bosch X. Primary Sjogren syndrome. BMJ. 2012 Jun 14;344:e3821. doi: 10.1136/bmj.e3821. No abstract available. PMID 22700787
- [Background] Danilovic A, Lucon AM, Srougi M, Shimizu MH, Ianhez LE, Nahas WC, Seguro AC. Protective effect of N-acetylcysteine on early outcomes of deceased renal transplantation. Transplant Proc. 2011 Jun;43(5):1443-9. doi: 10.1016/j.transproceed.2011.02.020. PMID 21693215
- [Derived] D'Agostino Gennari J, Deveza GBH, Ribeiro CT, Seguro AC, Aikawa NE, Shimizu MHM, Leon EP, Guedes LKN, Kupa LVK, Silva CAA, Bonfa E, Pasoto SG. Efficacy of N-acetylcysteine for treating dryness symptoms of Sjogren's disease: randomised placebo-controlled double-blind clinical study. Clin Exp Rheumatol. 2024 Dec;42(12):2427-2436. doi: 10.55563/clinexprheumatol/dmd5dv. Epub 2024 Sep 27. PMID 39360368